CLINICAL TRIAL: NCT05189509
Title: EXtending the tIme Window of Thrombolysis by ButyphThalide up to 6 Hours After Onset (EXIT-BT): a Prospective, Randomized, Blinded Assessment of Outcome and Open Label Multi-center Study
Brief Title: EXtending the tIme Window of Thrombolysis by ButyphThalide up to 6 Hours After Onset (EXIT-BT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: y (2021) 110
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — TNK-tissue plasminogen activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNK group (Experimental): intravenous thrombolysis with 0.25 mg/kg TNK, with the biggest dose of 25 mg
  Interventions: Drug: TNK-Tissue Plasminogen Activator
- control group (Placebo Comparator)
  Interventions: Drug: TNK-Tissue Plasminogen Activator

INTERVENTIONS:
Drug: TNK-Tissue Plasminogen Activator — 0.25 mg TNK thrombolysis

SUMMARY:
To date, the time window of intravenous thrombolysis is limited within 4.5 hours of stroke onset. Although EXTEND study has proved that intravenous thrombolysis can be extended from 4.5 to 9 hours, but the eligible patients must be selected by CTP. Thus, it is of clinical importance how to extend the time window of intravenous thrombolysis, which can benifit more patients. The current trial aims to investigate the effect of intravenous thrombolysis with TNK from 4.5 to 6 hours in ischemic stroke with help of Butyphthalide, which was found to be neuroprotective.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-80;
* ischemic stroke confirmed by brain CT or MRI
* the time from onset to treatment: 4.5-6 hours
* NIHSS≥4
* prestroke mRS≤1
* signed informed consent

Exclusion Criteria:

* prestroke mRS≥2
* planned endovascular treatment
* planned intravenous thrombolysis based on WAKE-UP or EXTEND study criterion
* any contraindiction of intravenous thrombolysis
* other unsuitable conditions judged by investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
symptomatic intracerebral hemorrhage | 36 hours
  any evidence of bleeding on the head CT scan associated with clinically significant neurological deterioration (NIHSS score ≥4 points increase)

SECONDARY OUTCOMES:
The proportion of excellent prognosis (mRS 0-1) | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome
The proportion of favourable prognosis (mRS 0-2) | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome
Distribution of modified Rankin Score | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome
Changes in National Institute of Health stroke scale (NIHSS) | 24 hours, 2 weeks
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
any intracerebral hemorrhage | 36 hours
  the evidence of bleeding on the head CT scan
any cerebral microbleeding(CMB) | 48 hours
  CMB is measured by SWI sequence
infarct volume | 48 hours
  infarct volume is measured by DWI sequence
proportion of death | Day 90
  death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen HS, Chen MR, Cui Y, Shen XY, Zhang H, Lu J, Zhao LW, Duan YJ, Li J, Wang YM, Min LQ, Zhao LH, Wan LS, Zhang ZH, Nguyen TN. Tenecteplase Plus Butyphthalide for Stroke Within 4.5-6 Hours of Onset (EXIT-BT): a Phase 2 Study. Transl Stroke Res. 2025 Jun;16(3):575-583. doi: 10.1007/s12975-024-01231-2. Epub 2024 Jan 19. PMID 38238620